CLINICAL TRIAL: NCT03208946
Title: Effects of a High Carboxymethyl-lysine (CML) Diet on Absorption and Excretion Levels in Healthy Adults
Brief Title: Effects of a High-CML Diet on Absorption and Excretion Levels in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Claudia Luévano-Contreras, Associate Professor, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CIBIUG-P32-2016
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Healthy
Keywords: Advanced glycation end products; Absorption; Excretion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-CML diet (Experimental): An isocaloric, high-CML content diet with a distribution of 55 to 63% carbohydrates, 12 to 15% protein, 25 to 30% lipids and less than 10% saturated fat.
  Interventions: Other: High-CML diet
- Low-CML diet (Sham Comparator): An isocaloric, low-CML content diet with a distribution of 55 to 63% carbohydrates, 12 to 15% protein, 25 to 30% lipids and less than 10% saturated fat.
  Interventions: Other: Low-CML diet

INTERVENTIONS:
Other: High-CML diet — Participants will be randomly assigned to either a high-CML or to a low-CML diet for 5 days, and they will receive the 5 corresponding meals (breakfast, lunch, snacks and dinner) during the 5 days of the intervention. These preparations will be elaborated by a catering company with indications and supervision by the research group. The intervention will be based on an isocaloric diet with a distribution of 55 to 63% carbohydrates, 12 to 15% protein, 25 to 30% lipids and less than 10% saturated fat and it macro and micronutrients will be similar in both diets. The only difference will be the CML content.
  Arms: High-CML diet
Other: Low-CML diet — Participants will be randomly assigned to either a high-CML or to a low-CML diet for 5 days, and they will receive the 5 corresponding meals (breakfast, lunch, snacks and dinner) during the 5 days of the intervention. These preparations will be elaborated by a catering company with indications and supervision by the research group. The intervention will be based on an isocaloric diet with a distribution of 55 to 63% carbohydrates, 12 to 15% protein, 25 to 30% lipids and less than 10% saturated fat and it macro and micronutrients will be similar in both diets. The only difference will be the CML content.
  Arms: Low-CML diet

SUMMARY:
The aim of this study is to evaluate the effect of carboxymethyl-lysine (CML) on the levels of absorption and excretion of CML, and in the microbiota of healthy adults. To achieve the objective, a randomized clinical trial will be carried out. Before the intervention, subjects will have a washout period for seven days, then they will be randomly assigned to either a high-CML or to a low-CML diet for 5 days. Both groups will consume the foods provided by the researchers at the research center. Diets for this intervention will be based on an isocaloric diet that will include breakfast, lunch, snacks and dinner.

Blood samples will be taken the first day, the second day of the intervention, and after the five days of the intervention. Urine and fecal samples will be taken the day before the intervention and after the intervention. CML levels will be measured by Liquid chromatography tandem-mass spectrometry in serum and urine samples to evaluate the levels of absorption and excretion. DNA extraction from the fecal sample will be carried out by a commercial kit. Bacterial log10 number of copies will be determined by using q-PCR.

DETAILED DESCRIPTION:
Advanced glycation end products (AGEs) are a heterogenous group of compounds form mainly by the Maillard reaction. AGEs can be found endogenously and in some foods. Several AGEs have been characterized, but carboxymethyl-lysine (CML) is one of the most widely studied in foods. Several studies have demonstrated the association between advanced glycation end products and several pathologies. However, few studies have focused on studying the absorption and excretion processes of these glycation products. Therefore, the objective of the study is to evaluate the effect of carboxymethyl-lysine (CML) on the levels of absorption and excretion of CML, and in the microbiota of healthy adults. To achieve the objective, a randomized clinical trial will be carried out, which will consist of a 7-day washout period during which participants will receive general recommendations that allow them to stick to a diet with a low CML content, adherence to these recommendations will be evaluated through three dietary records. At the end of the washing period, participants will be randomly assigned to either a high-CML or to a low-CML diet for 5 days. Participants will receive the 5 corresponding meals (breakfast, lunch, snacks and dinner) during the 5 days of the intervention, these preparations will be elaborated by a catering company with indications and supervision by the research group. Participants will assist to the research center to receive the breakfast, lunch and snacks. After lunch the subjects will receive a package containing a snack for mid-evening and the dinner. Adherence to the diet during the intervention period will be evaluated through a dietary record of foods.

The intervention will be based on an isocaloric diet with a distribution of 55 to 63% carbohydrates, 12 to 15% protein, 25 to 30% lipids and less than 10% saturated fat.

The diet with high content of CML will have twice the amount that the low diet, but with similar amounts of macro and micronutrients.

A blood sample will be taken on the first day of the intervention to measure CML basal levels. In order to evaluate the levels of CML absorption, the serum collection will be performed on the second day and at the end of the intervention. To evaluate the levels of CML excretion 24-hours urine will be collected the day before the intervention and the day after the dietary intervention finished. To evaluate the effects on the microbiota subjects will take a fecal sample the day before and a day after the intervention. Measurement of CML in serum, 24-hour urine and food will be performed by Liquid chromatography tandem-mass spectrometry. DNA extraction from the fecal sample will be carried out by a commercial kit. Bacterial log10 number of copies will be determined by using q-PCR.

ELIGIBILITY:
Inclusion Criteria:

* Adults 19 to 35 years old.
* Subjects with a body mass index (BMI) of 18.5 - 25 kg / m2
* Clinically healthy subjects, without presenting chronic diseases: diabetes mellitus, renal or cardiovascular disease.
* Non-smoking subjects.
* Subjects with low alcohol consumption.
* Subjects that do not consume food supplements.
* Subjects without known food allergies.
* Subjects without lactose intolerance or other foods.
* Subjects without gastrointestinal problems.
* Subjects who do not practice 150 minutes or more a week of physical exercise

Exclusion Criteria:

* Subjects with less than 80% adherence to the diet.
* Subjects who do not collect their indicated urine samples.
* Subjects presenting with an allergy, or adverse event during the intervention.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Serum levels of Carboxymethyl-lysine | six days
  Changes in serum levels of Carboxymethyl-lysine, a marker of AGEs, will be measured. Carboxymethyl-lysine serum levels will be measured by Liquid chromatography tandem-mass spectrometry.
Urinary levels of Carboxymethyl-lysine | six days
  Changes in urinary levels of Carboxymethyl-lysine, a marker of AGEs, will be measured. Carboxymethyl-lysine urinary levels will be measured by Liquid chromatography tandem-mass spectrometry.

SECONDARY OUTCOMES:
Bacterial log10 number of copies in fecal samples | six days
  Changes in bacterial log10 number of copies in fecal sample will be measured by qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: CLAUDIA LUEVANO CONTRERAS, PhD, Principal Investigator — Universidad de Guanajuato; Ma. Eugenia Garay-Sevilla, MD, Principal Investigator — Universidad de Guanajuato
Locations (1):
- University of Guanajuato, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No